CLINICAL TRIAL: NCT00604929
Title: The Effect of Carbohydrate and Protein Intake on Muscle Protein Synthesis During Endurance Exercise
Brief Title: Effect of Nutrition on Muscle Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Milou Beelen, Dr., Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC 83017
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: muscle protein synthesis; whole-body protein breakdown; nutrition
MeSH Terms: interventions — Carbohydrates; Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Dietary Supplement: carbohydrate and protein

INTERVENTIONS:
Dietary Supplement: carbohydrate and protein — The intake of carbohydrate and protein during endurance type exercise

SUMMARY:
The present proposal is designed to examine the effect of carbohydrate and protein co-ingestion on muscle protein synthesis during endurance type exercise activities. We hypothesize that muscle protein synthesis is higher when protein is co-ingested during exercise.

ELIGIBILITY:
Inclusion Criteria:

* recreationally endurance trained

Exclusion Criteria:

* BMI > 25 kg/m2
* Not physically active

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Differences in muscle protein synthesis rates between carbohydrate and carbohydrate + protein. | 1 day

SECONDARY OUTCOMES:
Difference in whole-body protein synthesis and breakdown between carbohydrate and carbohydrate plus protein. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: L van Loon, PhD, Principal Investigator — Maastricht University